CLINICAL TRIAL: NCT04734483
Title: The Effectiveness of Reconstructive Microsurgery on the Clinical and Functional State of Laryngeal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Astana Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aliya_Turayeva; dr.turayeva (Registry Identifier: Aliya Turayeva)
Record Dates: First submitted 2020-12-03; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Larynx Disease; Laryngeal Stenosis
Keywords: laryngeal stenosis; laryngeal MRI; laryngeal CT; pulmonary test; laryngoscopy
MeSH Terms: conditions — Laryngeal Diseases; Laryngostenosis | interventions — Spirometry; Magnetic Resonance Spectroscopy; Laryngoscopy; Neurofeedback

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, prospective, single-center
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- functional findings (Active Comparator): Participants with laryngeal stenosis
  Interventions: Diagnostic Test: spirometry
- to find anatomic feathers of larynx (Active Comparator): Participants with laryngeal stenosis
  Interventions: Radiation: MRI and CT; Other: Laryngoscopy
- to determine the type of stenosis of larynx and method of surgical treatment (Active Comparator): Participants with laryngeal stenosis
  Interventions: Diagnostic Test: spirometry; Radiation: MRI and CT; Other: Laryngoscopy; Other: electromyography
- determining the motor abilities of the muscles of the larynx (Active Comparator): Participants with laryngeal stenosis
  Interventions: Other: electromyography

INTERVENTIONS:
Diagnostic Test: spirometry — spirometry
  Arms: functional findings; to determine the type of stenosis of larynx and method of surgical treatment
Radiation: MRI and CT — MRI and CT
  Arms: to determine the type of stenosis of larynx and method of surgical treatment; to find anatomic feathers of larynx
Other: Laryngoscopy — laryngoscopy
  Arms: to determine the type of stenosis of larynx and method of surgical treatment; to find anatomic feathers of larynx
Other: electromyography — electromyography
  Arms: determining the motor abilities of the muscles of the larynx; to determine the type of stenosis of larynx and method of surgical treatment

SUMMARY:
To improve diagnostic methods for patients with laryngeal stenosis for the optimal determination of the technique of surgical treatment.

DETAILED DESCRIPTION:
The study include patients with laryngeal pathology in the otorhinolaryngology clinic of the 1-city hospital at Nur-Sultan city. All patients cheek up the necessary clinical, functional, diagnostic studies and treatment measures. It is planned to examine and operate on 70 patients with laryngeal pathology.

1. To study the features of the course of stenosis of the larynx under the influence of various factors, as well as traumatic injuries.
2. To develop optimal diagnostic methods for patients with laryngeal stenosis.
3. To assess the effectiveness of endolaryngeal microsurgery in patients with laryngeal stenosis.
4. To develop recommendations for the organization of treatment for stenosis of the larynx with an increase its functional state.

ELIGIBILITY:
Inclusion Criteria:

* medically diagnosed with stenosis of larynx
* patients who were observed larynx by MRI and CT
* patients who need surgical treatment of stenosis of larynx

Exclusion Criteria:

* pregnancy
* patients who has positive electromyography findings of motion of laryngeal muscles
* patients who has contraindications to surgical treatment on the other diseases
* patients who has not normal results of lab. analyses

Ages: 1 Year to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline forced expiratory volume | at baseline and at 24-week postrandomization
  Spirometry
Change from baseline area between vocal cords | at baseline and at 24-week postrandomization
  MRI and CT of larynx
Change from basiline vocal fold vibration | at baseline and at 24-week postrandomization
  Laryngoscopy and stroboscopy
Evaluate the motor system by recording action potential generated in muscle fibres like thyroarytenoid, lateral cricoarytenoid, posterior cricoarytenoid, interarytenoid, cricothyroid. | at baseline
  Electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Aliya Turayeva, PhD, Principal Investigator — Astana Medical Academy
Locations (2):
- Astana Medical University, Astana, Kazakhstan
- Saint-Petersburg Research Institute of Ear, Throat, Nose and Speech, Saint Petersburg, Russia